CLINICAL TRIAL: NCT06063759
Title: Comparative Measurement of Microcirculation and Other Parameters With the Vital USA VitalDetect™ in Patients With Diabetes Mellitus Type 1 and Type 2 Versus Healthy Paricipants
Brief Title: Comparative Measurement of Microcirculation and Other Parameters With the Vital USA VitalDetect™ in Patients With Diabetes Mellitus Type 1 and Type 2 Versus Healthy Participants
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was postponed due to manufacturing issues
Sponsor: Sciema UG (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: VIT-NGM-002
Record Dates: First submitted 2020-03-31; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: 3 groups with the same study procedures in sequential timely series.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VitalDetectTM (Other): Determination of microcirculating blood flow, glucose, SpO2, and heart rate.
  Interventions: Device: VitalDetect

INTERVENTIONS:
Device: VitalDetect — measurement of microcirculating blood flow, SpO2 (mmHg or %), heart rate (beats/min)

SUMMARY:
The purpose of this clinical study is to optimize the measurement algorithm of the Vital USA VitalDetectTM in measuring the microcirculating blood flow. Further optimization and finally the demonstration of the performance of the VitalDetectTM non-invasive monitoring biosensor in monitoring glucose, and heart rate in patients with type 1 and type 2 diabetes and healthy participants, when operated according to the instructions for use.

DETAILED DESCRIPTION:
The study procedures will be the same for all three groups during the single visit. In all groups of participants, the Vital USA VitalDetect™ will be individually introduced and assigned. During the experimental study visit, microcirculating blood flow (MBF), heart rate, and SpO2 will be measured using the Vital USA VitalDetect™ at 2 time points in between approx. 15 min. MBF will be measured in parallel by use of the LEA Medizintechnik O2C also using a finger on the same hand. The YSI glucose measurements will be employed to generate a robust algorithm for glucose measurements using the VitalDetect™. Parallel measurements of the heart rate and the SpO2 using a patient monitor (Edan iM8b) will be compared to the Vital USA VitalDetect™ device readings. Venous blood will be drawn from every subject to determine proinsulin, insulin and HbA1c values.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetic or healthy subject (25 Type 1, 25 Type 2, 50 healthy subjects)
* Subjects who are able to complete informed consent form (by him/herself or by his/her guardian);
* 18 years old and above;
* Anatomically suitable finger in discretion of the investigator

Exclusion Criteria:

* Does not meet inclusion criteria;
* Any conditions that may hamper good visual contact between the finger and sensor, such as raised birthmarks, scars, tattoos;
* Pregnancy;
* Nursing mothers;
* Any skin scratch(es), damage, over dry, long nails on the measured finger;
* Unsuitable finger with the device might be excluded if recognized during the trial;
* Medication containing nitrates

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-25 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the Vital USA VitalDetectTM for assessment of microcirculation (in AU) | 30 minutes
  Accuracy and performance of Vital USA VitalDetectTM for assessment of microcirculation (in AU) by measuring microcirculation using the VitalDetectTM in comparison to the LEA Medizintechnik O2C device.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Pfuetzner, MD, Principal Investigator — Pfützner Science & Health Institute GmbH
Locations (1):
- PSHI Praxis GmbH, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No